CLINICAL TRIAL: NCT04200313
Title: The Insulin-Only Bionic Pancreas Pivotal Trial: Testing the iLet in Adults and Children With Type 1 Diabetes
Brief Title: The Insulin-Only Bionic Pancreas Pivotal Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Beta Bionics, Inc. (Industry); Boston University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOBPPT; 1UC4DK108612-01 (NIH)
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes; Diabetes Mellitus, Type 1
Keywords: Artificial Pancreas; Closed-loop Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Bionic Pancreas (BP) (Experimental): Some adults and 1/2 peds will be randomized to use the Bionic Pancreas (BP) with lispro or aspart for 13 weeks
  Interventions: Combination Product: Bionic Pancreas (BP) with Aspart or Lispro
- Bionic Pancreas with Fiasp (BPFiasp) (Experimental): Some adults will be randomized to use the Bionic Pancreas (BP) with Fiasp for 13 weeks during RCT
  Interventions: Combination Product: Bionic Pancreas with Fiasp (BPFiasp)
- Usual Care (UC) (Other): Adults and peds will use their own diabetes insulin regimen plus continuous glucose monitoring (CGM) during the RCT
  Interventions: Other: Usual Care (UC)
- Bionic Pancreas Extension (Experimental): Used by all participants in the EXT study
  Interventions: Combination Product: Bionic Pancreas (BP) with Aspart or Lispro; Combination Product: Bionic Pancreas with Fiasp (BPFiasp)
- Transition Phase - BP Guidance (Experimental): Adults and peds will use their own diabetes insulin regimen plus SMBG and blinded continuous glucose monitoring (CGM) in the Transition phase and use dosing based on guidance from the BP system
  Interventions: Other: Usual Care (UC); Other: BP Guidance Insulin Dosing
- Transition- Pre-study dosing (Other): Adults and peds will use their own diabetes insulin regimen plus SMBG and blinded continuous glucose monitoring (CGM) in the Transition phase and use dosing based on their pre-study regimen
  Interventions: Other: Usual Care (UC)

INTERVENTIONS:
Combination Product: Bionic Pancreas (BP) with Aspart or Lispro — iLet Bionic Pancreas System, which consists of an integrated infusion pump, touchscreen display, Bluetooth radio, and insulin dosing algorithms, that automatically controls insulin delivery based on glucose values obtained by communicating with a Dexcom G6 sensor using lispro or aspart insulin.
  Other Names: iLet
  Arms: Bionic Pancreas (BP); Bionic Pancreas Extension
Combination Product: Bionic Pancreas with Fiasp (BPFiasp) — iLet Bionic Pancreas System, which consists of an integrated infusion pump, touchscreen display, Bluetooth radio, and insulin dosing algorithms, that automatically controls Fiasp insulin delivery based on glucose values obtained by communicating with a Dexcom G6 sensor.
  Arms: Bionic Pancreas Extension; Bionic Pancreas with Fiasp (BPFiasp)
Other: Usual Care (UC) — Using pre-study insulin regimen with the Dexcom G6 CGM
  Arms: Transition Phase - BP Guidance; Transition- Pre-study dosing; Usual Care (UC)
Other: BP Guidance Insulin Dosing — Pre-study insulin delivery method with SMBG and blinded CGM with dosing guidance by the BP
  Arms: Transition Phase - BP Guidance

SUMMARY:
This multi-center randomized control trial (RCT) will compare efficacy and safety endpoints using the insulin-only configuration of the iLet Bionic Pancreas (BP) System versus Usual Care (UC) during a 13-week study period. Participants may be enrolled initially into a screening protocol and then transfer into the RCT protocol, or they may enter directly into the RCT protocol. The RCT will be followed by an Extension Phase in which the RCT Usual Care (UC) Group will use the insulin-only configuration of the iLet Bionic Pancreas (BP) System for 3 months. At the completion of use of the BP system in the RCT only, participants will enter a 2-4 day Transition Phase and be randomly assigned to either transition back to their usual mode of therapy (MDI or pump therapy) based on therapeutic guidance from the iLet BP System or transition back to their usual mode of therapy based on what their own insulin regimens were prior to enrolling in the RCT.

There is an optional ancillary study to assess the safety of utilizing self-monitored blood glucose (SMBG) measurements instead of continuous glucose monitor (CGM) measurements as input into the iLet for ~48-60 hours. The Study is intended to mirror a real-world situation where CGM may not be available for an extended period of time (eg, user runs out of sensors and is awaiting new shipment).

DETAILED DESCRIPTION:
Primary Objective

• To compare the efficacy and safety of the insulin-only configuration of the iLet BP System (using insulin lispro, insulin aspart) the BP System using Fiasp (BPFiasp) [adults only]) in maintaining near-normal glycemia relative to usual care in a home-use study in adults and children with T1D.

Secondary Objectives • To assess the impact of the insulin-only configuration of the iLet BP System on quality of life and treatment satisfaction.

The study has four major parts: (1) the Test-Run Phase, (2) the RCT Period, (3) the Extension Phase for the UC Arm, and (4) the Transition Phase. These four parts are described below, and detailed in the main part of the protocol.

A Test-Run Phase will be conducted to (1) test the functionality of all aspects of the iLet BP System, (2) train the clinical staff on the execution of the clinical protocol, and (3) provide hands-on training with the device prior to initiating the RCT Period. The initial test run will be conducted at one site (MGH) with ~5 participants using the iLet BP system for 4-7 days. If there are no safety or consequential device issues, a test run will be conducted at each of the other 15 sites, with ~2 participants per site using the iLet BP system for 4-7 days. The iLet BP system will use insulin lispro or insulin aspart. Results of this Test-Run Phase will be evaluated for safety prior to beginning the RCT Period as described in section 3.3.

The 13-week, parallel-group, multi-center RCT Period is designed to compare the insulin-only iLet BP Group using insulin lispro, insulin aspart, or Fiasp (adults only); and a control group following usual care (UC Group). Upon completion of the RCT Period, the BP Group will enter the 2-4 day Transition Phase and the UC Group will enter the Extension Phase.

The UC Group Extension Phase will immediately follow the RCT Period. Participants from the UC Group who complete the primary outcome visit, miss no more than 3 of the maximum possible number of the weekly questionnaires, attend all clinic visits, and follow study procedures for collecting CGM data during the RCT Period, will be given the option to use the iLet BP system for 13 weeks. The visit schedule and procedures for the Extension Phase will be similar to that of the BP Group in the RCT Period.

A 2-4 day Transition Phase will be conducted for all participants who complete BP use at the end of the RCT Period (BP Group). Participants will be randomly assigned (1:1) to either transition back to their usual mode of therapy (MDI or pump therapy) based on therapeutic guidance from the iLet BP system or transition back to their usual mode of therapy based on what their own insulin regimens were prior to enrolling in the RCT Period. For those randomized to using their pre-study regimens, the dosing can be adjusted by the investigator to mitigate safety issues but should follow pre-study regimen as closely as possible.

An optional ancillary study will be offered to participants who are using the iLet at the time of the 13-week randomized trial visit. This will will assess the safety of utilizing blood glucose measurements instead of CGM measurements as input into the iLet for ~48-60 hours. It will be completed at the end of the RCT for those in the BP Group prior to the Transition Phase.

Test-Run Visit and Phone Contact Schedule

* Screening Visit - Eligibility assessed, informed consent, point-of-care/local HbA1c, testing and procedures similar to the RCT Screening Visit including psychosocial questionnaires; if eligible, BP system started.

  o For participants who completed the separate screening protocol, eligibility will be reassessed. Point-of-care/local HbA1c will be obtained if more than 28 days have elapsed. Participants will not need to repeat the psychosocial questionnaires.
* Phone contact after 1-2 days
* Shut-down visit at the end of the study period 4-7 days

RCT Period Visit and Phone Contact Schedule

* Screening Visit (which may be completed as part of a separate screening protocol)

  * Eligibility assessed, informed consent signed, point-of-care/local HbA1c, psychosocial questionnaires completed, blinded Dexcom G6 CGM sensor placed for non Dexcom G6 users.

    * For baseline data collection, participants using a personal Dexcom G6 who have at least 85% of possible glucose data in last 14 days can skip the blinded CGM wear
    * Participants using a personal Dexcom G6 with <85% of data will use their personal Dexcom G6.
    * For participants who completed the separate screening protocol, eligibility will be reassessed. Point-of-care/local HbA1c will be obtained if more than 28 days have elapsed. Participants will not need to repeat the psychosocial questionnaires or blinded CGM wear.
* If the separate screening protocol or Test Run Phase of this protocol was completed or blinded CGM wear is not needed, randomization can proceed immediately. If blinded CGM wear was performed as part of this protocol, randomization visit will occur14-21 days after screening.
* Prior to randomization, eligibility will be reassessed and blood drawn for central lab HbA1c
* BP study start/UC study start on day of Randomization Visit
* Phone contacts after 1-2 days and 7 (±2) days
* Visits at 2 weeks (±4 days), 6 weeks (±4 days), 10 weeks (±4 days), and ~13 weeks (91-98 days from randomization):

  * Participants in the UC Group will wear a blinded Dexcom G6 sensor throughout the entire study unless they are current users of the Dexcom G6 CGM, in which case they will continue to use their own Dexcom G6 CGM.
  * At the 6-week and 13-week visits, central lab HbA1c determination and psychosocial questionnaires

UC Group Extension Phase Visit and Phone Contact Schedule

* BP initiation at 13-week visit
* Phone contacts after 13 weeks plus 1-2 days and 14 weeks (±2 days)
* Visits at 15 weeks (± 4 days), 19 (±4 days), 23 (±4 days), and ~26 weeks (182-189 days):

  * At the 19-week and 26-week visits, central lab HbA1c determination and psychosocial questionnaires

Transition Phase Visit Schedule

* Randomization and transition to UC regimen at 13-week visit for RCT BP Group for a period of 2-4 days in duration.
* Visit ≤4 days later for end of study

Ancillary Study Day 1 (13-week visit of the RCT) - stop CGM, start blinded CGM, start SMBG at least every 2 hours during waking hours and at least once during each overnight for the next 48-60hrs.

Day 2: Phone call for safety

Day 3: stop iLet, stop blinded CGM, restart unblinded CGM, enter Transition Phase.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of T1D for at least one year and using insulin for at least 1 year 2. Diabetes managed using the same regimen (either pump or MDI, with or without CGM) for ≥ 3 months

  3. Age ≥ 6 years old
  * Exception: the initial 5-participant test run will be limited to >18 years old

    4. Current use of a CGM, or if not a CGM user, at least 3 blood glucose meter tests daily on average over the last 4 weeks (according to judgment of investigator if meter is not available).

    5. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial

    6. For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia.

    7. For participants >18 years old who live alone, participant has a relative or acquaintance who lives within 30 minutes of participant and is willing to be contacted to check on participant if study staff feel that participant may be experiencing a medical emergency and can't be reached.

    8. Investigator believes that the participant can safely use the iLet and will follow the protocol
  * The investigator will take into account the participant's HbA1c level, compliance with current diabetes management, and prior acute diabetic complications. For this reason, there is no upper limit on HbA1c specified for eligibility.

    9. If a GLP-1 agonist or pramlintide is being used, participant must be willing to discontinue use while the iLet BP system is being used, including the randomized trial and extension study.

Exclusion Criteria:

* Eligibility may be assessed initially in a separate screening protocol or at a screening visit in the RCT protocol. To be eligible for all phases of the study, a participant must meet all of the following inclusion criteria and none of the exclusion criteria:

Exclusion

1. Unable to provide informed consent (e.g. impaired cognition or judgment)
2. Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory)
3. Unable to speak and read English

   • For pediatric participants, both caregivers and participants must be able to speak and read English
4. Plan to change usual diabetes regimen in the next 3 months

   * This would include changing from MDI to pump. pump to MDI, change in insulin automation delivery system, starting a CGM if not previously used, changes in drug therapy specifically for glucose control except for changes in one insulin analog to another.
   * Changes in insulin dose, carb ratio, sensitivity factor and basal rate profile are allowed.
5. Current use of non-FDA approved closed-loop or hybrid closed-loop insulin delivery system
6. Use of Apidra as the pre-study rapid-acting insulin analog and unwilling to switch to lispro or aspart for the duration of the study
7. Known hemoglobinopathy (sickle cell trait is not an exclusion)
8. Current participation in another diabetes-related clinical trial
9. History of cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma, or history of complete pancreatectomy
10. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
11. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
12. Current use of SGLT2 inhibitors or a sulfonylurea drug (use more than 3 months prior to enrollment is acceptable)

    • If using GLP1 agonist, pramlintide, or metformin drugs must be on a stable dose for 3 months prior to enrollment (and as per inclusion criterion #8, must be willing to discontinue use of GLP-1 agonist or pramlintide while using the iLet BP system during the RCT and the extension phase).
13. Pregnant (positive urine hCG), breast feeding, plan to become pregnant in the next 3 months, or sexually active without use of contraception
14. For adults >18 years old, most recent (must be within the last 2 years) eGFR <30 ml/min OR currently in renal failure on dialysis

    • If no eGFR is available for an adult participant during the last 2 years, one must be obtained to confirm eligibility
15. Presence of a medical condition or use of a medication that, in the judgment of the investigator, clinical protocol chair, or medical monitor, could compromise the results of the study or the safety of the participant. Conditions to be considered by the investigator may include the following:

    * Alcohol or drug abuse
    * Use of prescription drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study
    * Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. climbing a flight of stairs) despite medical management, or within the last 12 months before screening a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
    * Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV
    * History of TIA or stroke in the last 12 months
    * Untreated or inadequately treated mental illness
    * History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
    * History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
16. Employed by, or having immediate family members employed by Beta Bionics, or being directly involved in conducting the clinical trial, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Paul Wadwa, MD, Principal Investigator — University of Colorado, Denver; Mark Daniels, MD, Principal Investigator — Children's Hospital of Orange County; Fran Cogen, MD, Principal Investigator — Children's National Research Institute; Keren Zhou, MD, Principal Investigator — The Cleveland Clinic; Andrew Muir, MD, Principal Investigator — Emory University; Davida Kruger, NP, Principal Investigator — Henry Ford Health System; Steven J Russell, MD, Principal Investigator — Massachusetts General Hospital; Robin Goland, MD, Principal Investigator — Naomi Berrie Center - Columbia University; Nelly Mauras, MD, Principal Investigator — Nemours Children's Health System; Bruce Buckingham, MD, Principal Investigator — Stanford University; Jeremy Pettus, MD, Principal Investigator — UC-San Diego; John Buse, MD, Principal Investigator — University of North Carolina, Chapel Hill; Irl Hirsch, MD, Principal Investigator — University of Washington; Jane Lynch, MD, Principal Investigator — UT Health Science Center - San Antonio; Perrin White, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Janet McGill, MD, Principal Investigator — Washington University School of Medicine; Jill Weissberg-Benchell, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Roy Beck, MD, PhD, Study Director — Jaeb Center for Health Research; Katrina Ruedy, MSPH, Study Director — Jaeb Center for Health Research; Philip Raskin, MD, Principal Investigator — UT Southwestern
Locations (16):
- United States (16):
  - Children's Hospital of Orange County (Pediatrics), Orange, California
  - University of California - San Diego (Adults), San Diego, California
  - Stanford University (Pediatrics and Adults), Stanford, California
  - Barbara Davis Center for Diabetes (Pediatrics and Adults), Aurora, Colorado
  - Children's National Health System (Pediatrics), Washington D.C., District of Columbia
  - Nemours Children's Clinic (Pediatrics), Jacksonville, Florida
  - Emory University (Pediatrics), Atlanta, Georgia
  - Massachusetts General Hospital - Diabetes Research Center (Peds and Adults), Boston, Massachusetts
  - Henry Ford Health System (Adults), Detroit, Michigan
  - Washington University (Adults), St Louis, Missouri
  - Naomi Berrie Diabetes Center at Columbia University (Pediatrics), New York, New York
  - University of Noth Carolina- Chapel Hill (Adults), Chapel Hill, North Carolina
  - Cleveland Clinic (Adults), Cleveland, Ohio
  - University of Texas- Southwestern (Pediatrics and Adults), Dallas, Texas
  - University of Texas Health Science Center (Pediatrics), San Antonio, Texas
  - University of Washington (Adults), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messer LH, Buckingham BA, Cogen F, Daniels M, Forlenza G, Jafri RZ, Mauras N, Muir A, Wadwa RP, White PC, Russell SJ, Damiano ER, El-Khatib FH, Ruedy KJ, Balliro CA, Li Z, Marak MC, Calhoun P, Beck RW. Positive Impact of the Bionic Pancreas on Diabetes Control in Youth 6-17 Years Old with Type 1 Diabetes: A Multicenter Randomized Trial. Diabetes Technol Ther. 2022 Oct;24(10):712-725. doi: 10.1089/dia.2022.0201.pub. PMID 36173237
- [Background] Mauras N, Damiano ER, El-Khatib FH, Marak MC, Calhoun P, Ruedy KJ, Balliro C, Li Z, Beck RW, Russell SJ. Utility and Safety of Backup Insulin Regimens Generated by the Bionic Pancreas: A Randomized Study. Diabetes Technol Ther. 2023 Jun;25(6):437-441. doi: 10.1089/dia.2022.0461. Epub 2023 Mar 22. PMID 36877259
- [Background] Li Z, Calhoun P, Ruedy KJ, Beck RW. Concordance of Central Laboratory Hemoglobin A1c Measurements from Capillary Kits Compared to Venous Draws in the Insulin-Only Bionic Pancreas Pivotal Trial. Diabetes Technol Ther. 2023 Jul;25(7):513-515. doi: 10.1089/dia.2023.0094. Epub 2023 May 2. PMID 37053531
- [Background] Kruger D, Kass A, Lonier J, Pettus J, Raskin P, Salam M, Trikudanathan S, Zhou K, Russell SJ, Damiano ER, El-Khatib FH, Ruedy KJ, Balliro C, Li Z, Marak MC, Calhoun P, Beck RW. A Multicenter Randomized Trial Evaluating the Insulin-Only Configuration of the Bionic Pancreas in Adults with Type 1 Diabetes. Diabetes Technol Ther. 2022 Oct;24(10):697-711. doi: 10.1089/dia.2022.0200. PMID 36173236
- [Background] Beck RW, Russell SJ, Damiano ER, El-Khatib FH, Ruedy KJ, Balliro C, Li Z, Calhoun P. A Multicenter Randomized Trial Evaluating Fast-Acting Insulin Aspart in the Bionic Pancreas in Adults with Type 1 Diabetes. Diabetes Technol Ther. 2022 Oct;24(10):681-696. doi: 10.1089/dia.2022.0167. PMID 36173235
- [Result] Bionic Pancreas Research Group; Russell SJ, Beck RW, Damiano ER, El-Khatib FH, Ruedy KJ, Balliro CA, Li Z, Calhoun P, Wadwa RP, Buckingham B, Zhou K, Daniels M, Raskin P, White PC, Lynch J, Pettus J, Hirsch IB, Goland R, Buse JB, Kruger D, Mauras N, Muir A, McGill JB, Cogen F, Weissberg-Benchell J, Sherwood JS, Castellanos LE, Hillard MA, Tuffaha M, Putman MS, Sands MY, Forlenza G, Slover R, Messer LH, Cobry E, Shah VN, Polsky S, Lal R, Ekhlaspour L, Hughes MS, Basina M, Hatipoglu B, Olansky L, Bhangoo A, Forghani N, Kashmiri H, Sutton F, Choudhary A, Penn J, Jafri R, Rayas M, Escaname E, Kerr C, Favela-Prezas R, Boeder S, Trikudanathan S, Williams KM, Leibel N, Kirkman MS, Bergamo K, Klein KR, Dostou JM, Machineni S, Young LA, Diner JC, Bhan A, Jones JK, Benson M, Bird K, Englert K, Permuy J, Cossen K, Felner E, Salam M, Silverstein JM, Adamson S, Cedeno A, Meighan S, Dauber A. Multicenter, Randomized Trial of a Bionic Pancreas in Type 1 Diabetes. N Engl J Med. 2022 Sep 29;387(13):1161-1172. doi: 10.1056/NEJMoa2205225. PMID 36170500
- [Derived] Shapiro JB, Vesco AT, Carroll MS, Weissberg-Benchell J. Psychometric Properties of the Automated Insulin Delivery: Benefits and Burdens Scale for Adults with Type 1 Diabetes. Diabetes Technol Ther. 2024 Nov;26(11):842-850. doi: 10.1089/dia.2024.0117. Epub 2024 May 31. PMID 38758212
- [Derived] Marak MC, Calhoun P, Damiano ER, Russell SJ, Ruedy KJ, Beck RW. Testing the Real-World Accuracy of the Dexcom G6 Pro CGM During the Insulin-Only Bionic Pancreas Pivotal Trial. Diabetes Technol Ther. 2023 Nov;25(11):817-821. doi: 10.1089/dia.2023.0287. Epub 2023 Oct 3. PMID 37668666
- [Derived] Weissberg-Benchell J, Vesco AT, Shapiro J, Calhoun P, Damiano ER, Russell SJ, Li Z, El-Khatib FH, Ruedy KJ, Balliro CA, Beck RW. Psychosocial Impact of the Insulin-Only iLet Bionic Pancreas for Adults, Youth, and Caregivers of Youth with Type 1 Diabetes. Diabetes Technol Ther. 2023 Oct;25(10):705-717. doi: 10.1089/dia.2023.0238. Epub 2023 Sep 5. PMID 37523175
- [Derived] Lynch J, Kanapka LG, Russell SJ, Damiano ER, El-Khatib FH, Ruedy KJ, Balliro C, Calhoun P, Beck RW. The Insulin-Only Bionic Pancreas Pivotal Trial Extension Study: A Multi-Center Single-Arm Evaluation of the Insulin-Only Configuration of the Bionic Pancreas in Adults and Youth with Type 1 Diabetes. Diabetes Technol Ther. 2022 Oct;24(10):726-736. doi: 10.1089/dia.2022.0341. PMID 36173238

RESULTS

PARTICIPANT FLOW:
Groups:
- Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L): Participants randomized to the Bionic Pancreas iLet with aspart/lispro insulin (BP-A/L) arm will use the iLet & Dexcom G6 CGM for 3 months
- Bionic Pancreas iLet With Fiasp Insulin (BP-F): Participants randomized to the Bionic Pancreas iLet with Fiasp insulin (BP-F) arm will use the iLet & Dexcom G6 CGM for 3 months
- Usual Care (UC): Participants randomized to Usual Care (UC) will continue using their usual insulin delivery method and a study CGM (Dexcom G6) for 3 months
- Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run): Upon completion of the RCT period, participants from the Bionic Pancreas iLet with Aspart/Lispro Insulin (BP-A/L) and Bionic Pancreas iLet with Fiasp Insulin (BP-F) groups voluntarily enrolled into the ancillary study testing iLet with inputted blood glucose measurements instead of CGM values for approximately 48 hours.
- Transition to Usual Care With Bionic Pancreas iLet Guidance (BP): Upon completion of either a) the RCT period for the Bionic Pancreas iLet with aspart/lispro insulin (BP-A/L) or Bionic Pancreas iLet with Fiasp insulin (BP-F) arms, or b) the Ancillary Study Testing iLet with Inputted Blood Glucose Measurements period, whichever is later, participants were randomized to transition back to their usual mode of therapy (MDI or pump therapy) based on therapeutic guidance from the iLet BP system.
- Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC): Upon completion of either a) the RCT period for the Bionic Pancreas iLet with aspart/lispro insulin (BP-A/L) or Bionic Pancreas iLet with Fiasp insulin (BP-F) arms, or b) the Ancillary Study Testing iLet with Inputted Blood Glucose Measurements period, whichever is later, participants were randomized to transition back to their usual mode of therapy (MDI or pump therapy) based on insulin regiments prior to enrolling in the RCT period.
- Usual Care Crossover to Bionic Pancreas iLet Extension (BPX): Upon completion of the RCT period for the Usual Care (UC) arm, select participants crossed over into the 3-month extension phase using the Bionic Pancreas with either Fiasp insulin or aspart/lispro insulin.
Period: RCT
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX)
Started | 219 | 114 | 107 | 0 | 0 | 0 | 0
Completed | 216 | 113 | 107 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 0 | 0 | 0 | 0 | 0
Period: BG Run Ancillary Study
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX)
Started | 0 | 0 | 0 | 58 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 54 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 0 | 0 | 0
Period: Transition Phase
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX)
Started | 0 | 0 | 0 | 0 | 148 | 149 | 0
Completed | 0 | 0 | 0 | 0 | 148 | 147 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0
Period: Extension Phase
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 90
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 84
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC) | Total
Number analyzed (Participants) | 219 | 114 | 107 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (19) | 42 (16) | 28 (20) | 32 (19)
Age, Customized [Count of Participants; unit: Participants]
  Age: <18 years | 112 | 0 | 53 | 165
  Age: ≥18 years | 107 | 114 | 54 | 275
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 62 | 41 | 210
  Male | 112 | 52 | 66 | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity Group: White Non-Hispanic | 157 | 98 | 83 | 338
  Race/Ethnicity Group: Black Non-Hispanic | 27 | 10 | 5 | 42
  Race/Ethnicity Group: Hispanic or Latino | 23 | 6 | 11 | 40
  Race/Ethnicity Group: Asian | 2 | 0 | 3 | 5
  Race/Ethnicity Group: American Indian/Alaskan Native | 1 | 0 | 1 | 2
  Race/Ethnicity Group: More than one race | 7 | 0 | 4 | 11
  Race/Ethnicity Group: Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 219 | 114 | 107 | 440
HbA1c [Mean (Standard Deviation); unit: %] | 7.9 (1.2) | 7.8 (1.2) | 7.7 (1.1) | 7.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: The primary outcome is superiority for central lab hemoglobin A1c at 13 weeks. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
mmol/mol | 56 (7.7) | 54 (6.6) | 61 (10.9)
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Non-inferiority for CGM-measured Time <54 mg/dL (Key Secondary Endpoint)
Description: The key secondary endpoint is CGM-measured time <54 mg/dL over 13 weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 0.33 [0.16 to 0.60] | 0.26 [0.12 to 0.48] | 0.24 [0.13 to 0.63]
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Non-Inferiority — Non-inferiority with a 1% non-inferiority margin; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Non-Inferiority — Non-inferiority with a 1% non-inferiority margin; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: CGM-measured Mean Glucose Level Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
mg/dL | 164 (15) | 155 (11) | 181 (32)
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: CGM-measured Percentage Time 70-180 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 65 (9) | 71 (8) | 54 (17)
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis

5. Secondary Outcome: CGM-measured Percentage Time >180 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 33 (9) | 27 (8) | 44 (18)
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis

6. Secondary Outcome: CGM-measured Percentage Time >250 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 8.5 [5.3 to 13.2] | 4.8 [2.7 to 7.6] | 14.9 [6.3 to 25.3]
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis

7. Secondary Outcome: CGM-measured Glucose Standard Deviation (SD) mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
mg/dL | 60 (11) | 52 (9) | 67 (16)
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p < 0.001, Mixed Models Analysis

8. Secondary Outcome: CGM-Measured Percentage Time <70 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 1.8 [1.1 to 2.9] | 1.7 [1.0 to 2.5] | 1.8 [0.8 to 3.1]
Statistical Analysis 1: Comparison: Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) vs Usual Care (UC); Test type: Superiority; p = 0.51, Mixed Models Analysis
Statistical Analysis 2: Comparison: Bionic Pancreas iLet With Fiasp Insulin (BP-F) vs Usual Care (UC); Test type: Superiority; p = 0.54, Mixed Models Analysis

9. Secondary Outcome: CGM-measured Percentage Time <54 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 0.33 [0.16 to 0.60] | 0.26 [0.12 to 0.48] | 0.24 [0.13 to 0.63]

10. Secondary Outcome: CGM-Measured Glucose Coefficient of Variation Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 36 (5) | 33 (4) | 37 (5)

11. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c <7.0%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c <7.0% at week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 65 | 49 | 27

12. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c <7.0% in Participants With Baseline HbA1c >7.5%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c <7.0% at week 13 in participants with baseline HbA1c >7.5%. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with a) non-missing central lab HbA1c measurements at randomization and at 13 weeks, and b) an HbA1c value >7.5% at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 115 | 60 | 56
Participants | 15 | 18 | 2

13. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c <7.5%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c <7.5% at week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 128 | 86 | 40

14. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c <8.0%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c <8.0% at week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 182 | 105 | 73

15. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c >9.0%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c >9.0% at week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 1 | 1 | 13

16. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c Improvement >0.5%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c improvement >0.5% from baseline to week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 100 | 62 | 13

17. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c Improvement >1.0%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c improvement >1.0% from baseline to week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 55 | 30 | 5

18. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c Relative Improvement >10%
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c relative improvement >10% from baseline to week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 72 | 42 | 5

19. Secondary Outcome: Other Secondary Efficacy Endpoint: HbA1c Improvement >1.0% or HbA1c <7.0% at 13 Weeks
Description: Other Secondary Efficacy Endpoint: Central lab hemoglobin A1c improvement >1.0% from baseline to week 13 or central lab hemoglobin A1c <7.0% at week 13. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with non-missing central lab HbA1c measurements at randomization and at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 108 | 66 | 30

20. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time in Range 70-140 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 39 (8) | 43 (7) | 33 (13)

21. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time in Range 70-120 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 23 (6) | 25 (6) | 21 (10)

22. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time <60 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 0.7 [0.4 to 1.1] | 0.5 [0.3 to 1.0] | 0.6 [0.3 to 1.3]

23. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Area Over the Curve 70 mg/dL Over 13 Weeks
Description: Area over the curve 70 mg/dL over the 13-week RCT period, measured as the mean of the differences between 70 mg/dL and CGM-measured glucose values below 70 mg/dL. For CGM-measured glucose values above 70 mg/dL, a value of 0 is used instead of the difference. For example, suppose a participant has 10 glucose readings of 78, 60, 59, 71, 80, 100, 110, 115, 120, and 118 mg/dL measured every 5 minutes. The distance between each reading below 70 mg/dL and 70 mg/dL is 0, 10, 11, 0, 0, 0, 0, 0, 0, and 0 mg/dL. The total area is 105 mg/dL*min; however, this value is then standardized by dividing by the length of time (50 min), resulting in a final CGM-measured area over the curve 70 mg/dL of 2.1 mg/dL.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
mg/dL | 0.18 [0.10 to 0.29] | 0.15 [0.08 to 0.25] | 0.16 [0.07 to 0.34]

24. Secondary Outcome: Other Secondary Efficacy Endpoint: Low Blood Glucose Index (LBGI)
Description: Other Secondary Efficacy Endpoint: CGM-measured low blood glucose index (LBGI) over 13 weeks. Ranges from 0 to 38.20, with higher values indicating more low CGM-measured glucose values over 13 weeks. Higher values are considered a worse outcome.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
units on a scale | 0.54 [0.38 to 0.76] | 0.55 [0.36 to 0.72] | 0.52 [0.31 to 0.88]

25. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Hypoglycemic Events
Description: Other Secondary Efficacy Endpoint: CGM-measured hypoglycemic event (at least 15 consecutive minutes with a sensor reading <54 mg/dL) rate over 13 weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Number of events per week
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Number of events per week | 0.68 [0.26 to 1.19] | 0.53 [0.24 to 1.10] | 0.48 [0.22 to 1.31]

26. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Hyperglycemic Events
Description: Other Secondary Efficacy Endpoint: CGM-measured hyperglycemic event (at least 90 minutes within a 120 minute period with a sensor reading >300 mg/dL) rate over 13 weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Number of events per week
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Number of events per week | 0.9 [0.4 to 2.0] | 0.4 [0.2 to 0.8] | 2.1 [0.6 to 4.2]

27. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time >300 mg/dL Over 13 Weeks
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Percentage | 2.4 [1.2 to 4.7] | 1.0 [0.4 to 1.9] | 6.0 [1.6 to 11.6]

28. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Area Under the Curve 180 mg/dL Over 13 Weeks
Description: Area under the curve 180 mg/dL over the 13-week RCT period, measured as the mean of the differences between 180 mg/dL and CGM-measured glucose values above 180 mg/dL. For CGM-measured glucose values under 180 mg/dL, a value of 0 is used instead of the difference. For example, suppose a participant has 10 glucose readings of 100, 120, 182, 200, 250, 193, 179, 150, 140 and 118 mg/dL measured every 5 minutes. The distance between each reading above 180 mg/dL and 180 mg/dL is 0, 0, 2, 20, 70, 13, 0, 0, 0, and 0 mg/dL. The total area is 525 mg/dL*min; however, this value is then standardized by dividing by the length of time (50 min), resulting in a final CGM-measured area under the curve 180 mg/dL of 10.5 mg/dL.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
mg/dL | 17.2 [11.5 to 23.1] | 10.8 [8.1 to 15.4] | 26.2 [13.1 to 42.2]

29. Secondary Outcome: Other Secondary Efficacy Endpoint: High Blood Glucose Index (HBGI)
Description: Other Secondary Efficacy Endpoint: CGM-measured high blood glucose index (HBGI) over 13 weeks. Ranges from 0 to 57.27, with higher values indicating more high CGM-measured glucose values over 13 weeks. Higher values are considered a worse outcome.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
units on a scale | 7.4 [5.9 to 9.1] | 5.8 [4.8 to 6.9] | 10.0 [6.4 to 14.3]

30. Secondary Outcome: Other Secondary Efficacy Endpoint: Mean of Daily Difference in Mean Glucose
Description: Other Secondary Efficacy Endpoint: CGM-measured mean of daily difference in mean glucose over 13 weeks
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
mg/dL | 20 (7) | 16 (5) | 30 (11)

31. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time in Range 70-180 mg/dL >70% Over 13 Weeks
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 56 | 65 | 23

32. Secondary Outcome: Other Secondary Efficacy Endpoint: Time in Range 70-180 mg/dL Improvement From Baseline to 13 Weeks ≥5%
Description: Other Secondary Efficacy Endpoint: CGM-measured percentage time in range 70-180 mg/dL improvement from baseline to 13 weeks ≥5%
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 159 | 90 | 55

33. Secondary Outcome: Other Secondary Efficacy Endpoint: Time in Range 70-180 mg/dL Improvement From Baseline to 13 Weeks ≥10%
Description: Other Secondary Efficacy Endpoint: CGM-measured percentage time in range 70-180 mg/dL improvement from baseline to 13 weeks ≥10%
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 146 | 84 | 43

34. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time <70 mg/dL <4%
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 194 | 109 | 86

35. Secondary Outcome: Other Secondary Efficacy Endpoint: CGM-measured Percentage Time <54 mg/dL <1%
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 190 | 108 | 88

36. Secondary Outcome: Other Secondary Efficacy Endpoint: Blood Glucose Risk Index (LBGI + HBGI)
Description: Other Secondary Efficacy Endpoint: CGM-measured Blood Glucose Risk Index (LBGI + HBGI) over 13 weeks. Calculated as Low Blood Glucose Index (LBGI) + High Blood Glucose Index (HBGI). Ranges from 0 to 57.27, with higher values indicating more low or high CGM-measured glucose values over 13 weeks. Higher values are considered a worse outcome. LBGI and HBGI are inversely related: the presence of a high CGM-measured glucose reading removes an opportunity for a low glucose reading to exist and vice versa, therefore a maximum HBGI of 57.27 and a maximum LGBI of 38.20 cannot exist simultaneously. For instance, if a participant had glucose values of only 401 mg/dL, then the participant has no low glucose values, and therefore their HBGI = 57.27 and LBGI = 0. If a participant had only glucose values of 39 mg/dL, then the participant has no high glucose values, and therefore their HBGI = 0 and LBGI = 38.20. Consequently, the maximum blood glucose risk index is 57.27.
Time Frame: 13 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
units on a scale | 8.0 [6.7 to 9.7] | 6.3 [5.3 to 7.5] | 10.7 [6.9 to 14.9]

37. Secondary Outcome: Other Secondary Efficacy Endpoint: Improvement in HbA1c > 0.5% Without an Increase in Time < 54 mg/dl by > 0.5% OR Improvement in Time < 54 mg/dl by > 0.5% Without an Increase in HbA1c by > 0.5%
Description: Other Secondary Efficacy Endpoint: Baseline to week 13 improvement in central lab hemoglobin A1c >0.5% without an increase in CGM-measured percentage time <54 mg/dl by >0.5% OR improvement in CGM-measured percentage time <54 mg/dl by >0.5% without an increase in central lab hemoglobin A1c by >0.5%. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Population: Only including participants with a) at least 168 hours of CGM data at baseline and over the 13-week follow-up period, and b) non-missing central lab HbA1c measurements at randomization and week 13.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 103
Participants | 104 | 62 | 15

38. Secondary Outcome: Other Secondary Efficacy Endpoint: Improvement in Time 70-180 mg/dl by >10% Without an Increase in Time < 54 mg/dl by > 0.5% OR Improvement in Time < 54 mg/dl by > 0.5% Without a Decrease in Time 70-180 mg/dl by > 10%
Description: Other Secondary Efficacy Endpoint: Baseline to 13-week improvement in CGM-measured percentage time 70-180 mg/dL by >10% without an increase in CGM-measured percentage time <54 mg/dL by >0.5% OR improvement in CGM-measured percentage time <54 mg/dL by >0.5% without a decrease in CGM-measured percentage time 70-180 mg/dL by >10%
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 120 | 74 | 25

39. Secondary Outcome: Other Secondary Efficacy Endpoint: Mean Glucose <154 mg/dL and Time <54 mg/dL <1%
Description: Other Secondary Efficacy Endpoint: CGM-measured mean glucose <154 mg/dL and percentage time <54 mg/dL <1% over 13 weeks
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 46 | 51 | 17

40. Secondary Outcome: Other Secondary Efficacy Endpoint: Time in Range 70-180 mg/dL >70% and Time <54 mg/dL <1%
Description: Other Secondary Efficacy Endpoint: CGM-measured percentage time in range 70-180 mg/dL >70% and percentage time <54 mg/dL <1% over 13 weeks
Time Frame: 13 weeks
Population: Only including participants with at least 168 hours of CGM data at baseline and over the 13-week follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 218 | 113 | 107
Participants | 52 | 63 | 16

41. Secondary Outcome: Other Secondary Efficacy Endpoint: Total Daily Insulin (Units/kg)
Description: Other Secondary Efficacy Endpoint: Total daily insulin (units/kg) from week 13 site-reported insulin data for the UC group and iLet pump device data over 13 weeks for the BP-A/L and BP-F groups.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Insulin units per kg
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 217 | 110 | 107
Insulin units per kg | 0.86 (0.33) | 0.65 (0.19) | 0.81 (0.34)

42. Secondary Outcome: Other Secondary Efficacy Endpoint: Percentage Change in the TDD of Insulin Over the First Two-week Period Relative to the TDD of Insulin in the Last Two-week Period
Description: Other Secondary Efficacy Endpoint: Percentage change in the TDD of insulin over the first two-week period relative to the TDD of insulin in the last two-week period from iLet pump device data over 13 weeks for the BP-A/L and BP-F groups.
Time Frame: Weeks 1-2 and weeks 12-13
Population: iLet pump device was given to BP-A/L and BP/F groups only.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F)
Number analyzed (Participants) | 202 | 107
Percentage change | 5 (21) | 6 (26)

43. Secondary Outcome: Other Secondary Efficacy Endpoint: Body Weight at Week 13
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 215 | 113 | 107
kg | 69 (24) | 84 (19) | 70 (27)

44. Secondary Outcome: Other Secondary Efficacy Endpoint: Body Mass Index (BMI) at Week 13
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 211 | 105 | 102
kg/m^2 | 25.5 (6.3) | 29.2 (5.5) | 25.2 (7.5)

45. Secondary Outcome: Other Secondary Efficacy Endpoint: Mean Participant-reported Number of Hypoglycemic Events Requiring Carbohydrate Treatment Per 24 Hours
Description: Mean participant-reported number of hypoglycemic events requiring carbohydrate treatment per 24 hours, based on the responses to the question, 'How many times in the last 24 hours did you take carbohydrates to treat a low blood sugar?' administered to participants once weekly during the 13-week RCT period.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Number of events in last 24 hours
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 217 | 108 | 106
Number of events in last 24 hours | 1.0 (0.7) | 0.9 (0.7) | 0.8 (0.6)

46. Secondary Outcome: Other Secondary Efficacy Endpoint: Mean Participant-reported Grams of Carbohydrate Taken Specifically to Prevent or Treat Hypoglycemic Events Per 24 Hours
Description: Mean participant-reported number of hypoglycemic events requiring carbohydrate treatment per 24 hours, based on the responses to the question, 'Estimate the total amount of grams of carbohydrates you were given to treat these low blood sugars', which is a follow-up question to 'How many times in the last 24 hours did you take carbohydrates to treat a low blood sugar?'. Both questions were administered to participants once weekly during the 13-week RCT period.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: grams in last 24 hours
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 217 | 108 | 106
grams in last 24 hours | 12.7 (10.1) | 12.6 (12.0) | 12.5 (8.8)

47. Other Pre Specified Outcome: Safety Outcome Measure: Severe Hypoglycemia Events
Description: Safety Outcome Measure: Severe hypoglycemia (SH) events with cognitive impairment requiring assistance of a third party for treatment.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Participants | 10 | 3 | 2

48. Other Pre Specified Outcome: Safety Outcome Measure: Diabetic Ketoacidosis Events
Description: Safety Outcome Measure: Diabetic ketoacidosis events (DKA) over 13 weeks as defined by the Diabetes Control and Complications Trial: symptoms such as polyuria, polydipsia, nausea, or vomiting; serum ketones >1.5 mmol/L or large/moderate urine ketones; either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate <15; and treatment provided in a health care facility.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Participants | 0 | 2 | 0

49. Other Pre Specified Outcome: Safety Outcome Measure: Other Serious Adverse Events
Description: Safety Outcome Measure: Serious adverse events excluding SH and DKA
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 219 | 114 | 107
Participants | 3 | 0 | 2

50. Other Pre Specified Outcome: Safety Outcome Measure: Worsening of HbA1c by >0.5%
Description: Safety Outcome Measure: Worsening of central lab hemoglobin A1c from baseline to week 13 by >0.5%. Glycated Hemoglobin A1C (HbA1c) is a physiological marker of the percentage of red blood cells that have glycated (bonded with a sugar). HbA1c is used to measure changes in average blood sugar over the past three months.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC)
Number analyzed (Participants) | 212 | 111 | 104
Participants | 17 | 7 | 8

ADVERSE EVENTS:
Time Frame: From protocol entry through last study date, which is approximately 13 weeks per participant with an additional 13 weeks (i.e. weeks 14-26) for BPX participants only.
Arm/Group | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) | Usual Care (UC) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX)
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/114 | 0/107 | 0/58 | 0/148 | 0/149 | 0/90
Serious Adverse Events (participants affected / at risk) | 13/219 | 5/114 | 4/107 | 0/58 | 0/148 | 0/149 | 3/90
Other Adverse Events (participants affected / at risk) | 119/219 | 57/114 | 4/107 | 2/58 | 4/148 | 3/149 | 43/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) (N=219) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) (N=114) | Usual Care (UC) (N=107) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) (N=58) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) (N=148) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) (N=149) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX) (N=90)
Severe Hypoglycemia (Endocrine disorders) | 10 (10) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attempted suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Primary spontaneous pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bionic Pancreas iLet With Aspart/Lispro Insulin (BP-A/L) (N=219) | Bionic Pancreas iLet With Fiasp Insulin (BP-F) (N=114) | Usual Care (UC) (N=107) | Bionic Pancreas iLet With Inputted Blood Glucose Measurements Run-In (BG Run) (N=58) | Transition to Usual Care With Bionic Pancreas iLet Guidance (BP) (N=148) | Transition to Usual Care Without Bionic Pancreas iLet Guidance (UC) (N=149) | Usual Care Crossover to Bionic Pancreas iLet Extension (BPX) (N=90)
Hyperglycemia or ketosis events without meeting criteria for diabetic ketoacidosis (Endocrine disorders) | 111 (214) | 50 (66) | 1 (2) | 2 (2) | 4 (4) | 3 (3) | 41 (81)
Hypoglycemia (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter infection (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrown toe nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leg fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (8):
  • Study Protocol (2021-04-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/Prot_010.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/SAP_011.pdf
  • Informed Consent Form: RCT ICF (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/ICF_004.pdf
  • Informed Consent Form: RCT Assent (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/ICF_005.pdf
  • Informed Consent Form: BG Run iLet Ancillary Study ICF (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/ICF_006.pdf
  • Informed Consent Form: BG Run iLet Ancillary Study Assent (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/ICF_007.pdf
  • Informed Consent Form: Screening ICF and Assent (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/ICF_008.pdf
  • Informed Consent Form: Test Run ICF and Assent (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT04200313/ICF_009.pdf